CLINICAL TRIAL: NCT03950700
Title: Bupivacaine in the Treatment of Postoperative Pain of Impacted Third Molar Extraction. A Randomized Clinical Trial.
Brief Title: Bupivacaine in the Treatment of Postoperative Pain of Impacted Third Molar Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Pablo Correa, Chief of Posgraduates Programs of Dentistry, CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 791
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Teeth, Impacted
Keywords: Analgesia; Bupivacaine; Postoperative pain; Third molar; Extraction
MeSH Terms: conditions — Tooth, Impacted; Agnosia; Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: In all patients, both impacted lower third molars are surgically removed in one session, beginning the extractions in the right side. Subsequently, one of the alveolus will be irrigated with 4ml of bupivacaine 0.5% with adrenaline vasoconstrictor 1: 200,000 (BUPIROP® 0.5% ROPSOHN® THERAPEUTICS SAS), the contralateral alveolus will be irrigated with 4 ml of saline solution 0.9% (Baxter laboratories) prior to the placement of the suture for the closure of the surgical wound, using the aspiration to avoid the exit of the medication out of the alveolus.
Who Masked: Participant
Masking Description: The decision to use another substance for the irrigation of the alveolus will be taken in a randomized manner.Through numerical assignment according to the order of surgical scheduling. The patients with even numbers are irrigated on the right side with bupivacaine and on the left side with saline. Patients with odd numbers will be irrigated in the opposite way.
  Patients will be considered blinded to the drug of choice, and they will not know what type of solution will be administered on each side.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine solution (Experimental): In all patients, both impacted lower third molars are surgically removed in one session, beginning the extractions in the right side. Subsequently, one of the alveolus will be irrigated with 4ml of bupivacaine 0.5% with adrenaline vasoconstrictor 1: 200,000 (BUPIROP® 0.5% ROPSOHN THERAPEUTICS SAS), the contralateral alveolus will be irrigated with 4 ml of saline solution 0.9% (Baxter laboratories) prior to the placement of the suture for the closure of the surgical wound, using the aspiration to avoid the exit of the medication out of the alveolus.
  Interventions: Drug: Bupivacaine-epinephrine
- Saline solution (Placebo Comparator): In all patients, both impacted lower third molars are surgically removed in one session, beginning the extractions in the right side. Subsequently, one of the alveolus will be irrigated with 4ml of bupivacaine 0.5% with adrenaline vasoconstrictor 1: 200,000 (BUPIROP® 0.5% ROPSOHN THERAPEUTICS SAS), the contralateral alveolus will be irrigated with 4 ml of saline solution 0.9% (Baxter laboratories) prior to the placement of the suture for the closure of the surgical wound, using the aspiration to avoid the exit of the medication out of the alveolus.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — BUPIROP® 0.5% ROPSOHN THERAPEUTICS S.A.S
  Other Names: Bupivacaine 0.5% with adrenaline vasoconstrictor 1: 200,000
  Arms: Bupivacaine solution
Drug: Saline Solution — Saline solution 0.9% (Baxter laboratories).
  Other Names: Saline solution 0.9%
  Arms: Saline solution

SUMMARY:
The third molars are the teeth that are most frequently included and impacted, extraction is one of the most performed treatments by maxillofacial surgeons in their clinical practice. Its surgical extraction is accompanied by an inflammatory process, which generates pain, edema and trismus. The use of alternatives that offer prolonged analgesia, like the use of bupivacaine, reduce the pain of the patient after an extraction of third molars, allows the reduction of morbidity and the rapid return to daily activities.

In addition, it allows a better experience in the dental consultation.

Investigators hypothesis is:

Irrigation of the alveolus with 4 ml of 0.5% bupivacaine is effective for the reduction of post-operative pain in extraction of impacted lower third molars

DETAILED DESCRIPTION:
Clinical, randomized, experimental, single blind study. The sample for the present study will consist of 40 patients who attend consecutively to maxillofacial surgery, to perform third molar surgical extraction.

The sample size defined for the present study is 40 patients, each with two extractions of third molars for a total of 80 extractions that will be randomized in each patient for the treatment of Bupivacaine and saline respectively.

For the calculation of statistical power with the sample size previously defined to compare the postoperative pain level 4, 12 and 24 hours after the extraction of lower third molars in two groups (Bupivacaine and saline).

With the sample size, investigators defined, calculated, statistical power, test and use, comparison, pain levels, at 4 and 12 hours, with a power greater than 90%. The study will have sufficient power for the study to be conclusive, regardless of whether it finds statistically significant differences or not.

The surgical procedure will be performed by a single oral and maxillofacial surgeon, following the same surgical technique for the extraction of impacted molars, in all patients, including the sulcular flap up to the second molar, with a posterior complementary incision of 45 degrees, without anterior incision Complementary. The osteotomy is performed with a high speed carbide surgical bur. The patients will not receive a previous medication.

In all patients, both impacted lower third molars are surgically removed in one session, beginning the extractions in the right side. Subsequently, one of the alveolus will be irrigated with 4ml of bupivacaine 0.5% with adrenaline vasoconstrictor 1: 200,000 (BUPIROP® 0.5%), the contralateral alveolus will be irrigated with 4 ml of saline solution 0.9% (Baxter laboratories) prior to the placement of the suture for the closure of the surgical wound, using the aspiration to avoid the exit of the medication out of the alveolus.

The decision to use another substance for the irrigation of the alveolus will be taken in a randomized manner.Through numerical assignment according to the order of surgical scheduling. The patients with even numbers are irrigated on the right side with bupivacaine and on the left side with saline. Patients with odd numbers will be irrigated in the opposite way.

Before starting the surgical procedure, the disposable syringes will be marked with their respective content, either bupivacaine 0.5% or saline solution 0.9%, each with 4 ml of the medication.

Patients will be considered blinded to the drug of choice, and patients will not know what type of solution will be administered on each side.

All patients will be medicated with: amoxicillin 500mg every 6 hours for 7 days, acetaminophen 500mg every 6 hours for 5 days, and ibuprofen 400mg every 6 hours for 5 days.

Postoperative pain will be evaluated at 4, 12 and 24 hours after surgery, using the pain visual analog scale from 1 to 10, by telephone call. Patients will be instructed to rate their pain intensity on each side from one to ten.

The information collected in the form will be digitized in a spreadsheet in Excel, to be analyzed in the program IBM® SPSS® version 21. All independent quantitative variables will be summarized by descriptive statistics (average or median, standard deviation o Interquartile range), while qualitative variables will be described with proportions. To compare the pain levels between the two treatments at 4, 12 and 24 hours, the Student's t-test for independent samples or, failing that, the Mann-Whitney U-test will be used.

Prior to this analysis, the normality of the postoperative pain variable (analogous visual scale) will be assessed using the Shapiro Wilk test. A level of significance of 5% will always be assumed for the contrasting statistical tests.

The univariate descriptive analysis will be presented through a summary table. In addition, an error bar graph will be used to show the levels of postoperative pain for each treatment at 4, 12 and 24 hours.

The clinical trial embraces the Declaration of Helsinki of ethical principles for medical research in humans.

Prior to carrying out the study, each of the participants will be explained what the research consists of, participants will be informed about possible adverse reactions to the local anesthetic Bupivacaine, such as drug reaction, altered blood pressure and heart rate, nausea. , vomiting, headaches and allergic skin reactions. At all times there will be a diligent management of the therapy and close observation establish the rules for the handling of personal data in clinical history.

An informed consent will be given to each patient, who will read and explain what is stipulated in it before consenting, to ensure that the participant who signs the informed consent agrees to perform the procedure as stipulated in the statement of the investigation.

The privacy of the individual, subject of investigation, will be protected, identifying it only when the results require it and this authorizes it.

The investigation will be suspended immediately, upon noticing any risk or damage to the health of the subject in whom the investigation is carried out.

ELIGIBILITY:
Inclusion Criteria:

* Lower third molars impacted bilaterally requiring an osteotomy for their extraction and which are located spatially within the following positions or classes according to Pell & Gregory (1933).

  * Position B (occlusal plane of the impacted tooth between the occlusal plane and the cervical line of the second molar).
  * Position C (tooth impacted below the cervical line of the second molar).
  * Class II (space between the second molar and the mandibular branch smaller than the distal mesial diameter of the third molar).
  * Class III (All or most of the third molar is inside the mandibular branch).
* Systemically healthy patients (ASA I-II).

Exclusion Criteria:

We exclude patients who present a history of infectious processes in the abscess area of third molars or who, for medical reasons, chronically use some type of analgesia.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity Measure: pain visual analog scale | 4, 12 and 24 postoperative hours
  To identify the analgesia obtained with the alveolus irrigation with bupivacaine at 4, 12 and 24 postoperative hours, by applying the analogous visual pain scale in each third molar object of study.
  Postoperative pain will be evaluated at 4, 12 and 24 hours after surgery, using the Likert pain visual analog scale from 1 to 10. There being 1 absence of pain and 10 the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Emilio Correa Echeverri, Principal Investigator — CES University
Locations (1):
- CES University, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No
The disclosure of the data obtained in this study will be made through the publication of the trial in a scientific journal

REFERENCES:
- [Result] Khorshidi Khiavi R, Pourallahverdi M, Pourallahverdi A, Ghorani Khiavi S, Ghertasi Oskouei S, Mokhtari H. Pain control following impacted third molar surgery with bupivacaine irrigation of tooth socket: a prospective study. J Dent Res Dent Clin Dent Prospects. 2010 Fall;4(4):105-9. doi: 10.5681/joddd.2010.027. Epub 2010 Dec 21. PMID 23346335
- [Result] Brajkovic D, Biocanin V, Milic M, Vucetic M, Petrovic R, Brkovic B. Quality of analgesia after lower third molar surgery: A randomised, double-blind study of levobupivacaine, bupivacaine and lidocaine with epinephrine. Vojnosanit Pregl. 2015 Jan;72(1):50-6. doi: 10.2298/vsp1501050b. PMID 26043591